CLINICAL TRIAL: NCT02310919
Title: Concomitant Administration of FSH With a Low Dose of hCG (1,500 IU) Has Equivalent Oocyte Developmental Competence While Decreasing the Exposure to hCG in IVF Cycles: A Double Blind Randomized Control Trial
Brief Title: Administration of Follicle-stimulating Hormone (FSH) and Low Dose Human Chorionic Gonadotropin (hCG) for Oocyte Maturity While Decreasing hCG Exposure in In Vitro Fertilization (IVF) Cycles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P0503461
Record Dates: First submitted 2014-09-04; First posted 2014-12-08 (Estimated); Results first posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Infertility
Keywords: Infertility; In vitro fertilization; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose hCG plus FSH co-trigger (Experimental): On the day of ovulation trigger the patient will receive hCG 1,500 IU SQ plus FSH 450 IU SQ
  Interventions: Drug: Low dose hCG plus FSH co-trigger
- Standard dose of hCG alone (Active Comparator): On the day of ovulation trigger the patient will receive standard dose of hCG (10,000 or 5,000 IU SQ)
  Interventions: Drug: Standard dose of hCG

INTERVENTIONS:
Drug: Low dose hCG plus FSH co-trigger — Low dose hCG (1,500 IU) plus FSH (450 IU) co-trigger
  Arms: Low dose hCG plus FSH co-trigger
Drug: Standard dose of hCG — Standard dose of hCG (10,000 or 5,000 IU) trigger
  Arms: Standard dose of hCG alone

SUMMARY:
This is a randomized, double-blind, single center clinical trial study to compare oocyte competence and risk of ovarian hyperstimulation syndrome (OHSS) after receiving the standard dose of human chorionic gonadotropin (hCG) ovulation trigger or a lower dose of hCG plus concomitant follicle stimulating hormone (FSH) co-trigger in women undergoing in vitro fertilization (IVF).

DETAILED DESCRIPTION:
The success rate of assisted reproductive technology (ART) has dramatically increased due to the improvements in embryo culture, laboratory conditions, and optimization of different ovarian stimulation protocols. Recent data shows that if hCG is not administered for oocyte maturation, severe OHSS is very rare. However, with gonadotropin releasing hormone (GnRH) agonist cycles, hCG is required. Previous studies have revealed that a smaller dose of hCG used for ovulation trigger versus the standard dose can have the same effect on the induction of final oocyte maturation and can possibly reduce the risk of OHSS . However, the minimal dose required of hCG to maintain maximal success rates of IVF is not known as it has not been adequately studied in randomized controlled trials. Interestingly, our previous randomized controlled study revealed that concomitant administration of FSH and hCG (10,000 IU), a more physiological process, improved developmental oocyte competence. In that study, there was no OHSS in the group that received the FSH co-trigger. A subsequent study performed a randomized trial to determine if FSH co-trigger reduced the incidence of OHSS and found that, it may prevent OHSS. Additionally, our own clinical experience (unpublished data) reveals that administering 1,500 IU hCG plus 450 IU FSH co-trigger is enough to promote adequate (i.e. non-inferior) oocyte maturation while not increasing the risk of developing OHSS in high risk patients. Given these findings, we propose a further modification of ovulation trigger with decreased exposure to hCG. Our objective is to determine if concomitant administration of FSH with a decreased dose of hCG versus a standard dose of hCG alone for ovulation will promote adequate oocyte maturation and quality, while decreasing the risk of OHSS. The selected FSH dose of 450 IU is thought to parallel the physiologic FSH surge observed in a natural cycle. We have chosen 1,500 IU as the designated low dose of hCG based on previous studies showing that even hCG doses as low as 2,000 IU allows oocytes to undergo maturation as well as our own clinical experience that has demonstrated adequate oocyte maturity and fertilization in patients chosen to receive 1,500 IU of hCG, due to the risk of OHSS.

Study participants will be recruited from the Reproductive Endocrinology and Infertility Clinic at University of California at San Francisco Center for Reproductive Health. Couples undergoing IVF will be offered participation in the study.

Approximately 100 subjects will be randomized at the time of enrollment to receive either the standard dose of hCG alone or low dose hCG (1,500 IU) + FSH (450 IU) for oocyte maturation trigger by the research coordinator. There will be about 50 subjects in each study arm.

Each subject will undergo a standard IVF stimulation protocol chosen by their primary physician. Study participants will receive a syringe (prepared by the research coordinator) on the day of ovulation trigger containing either the standard dose of hCG or low dose hCG + FSH according to the randomization. The subjects will be triggered with the following:

1. Control arm: Standard dose of hCG (10,000 or 5,000 IU) or
2. Experimental arm: hCG 1,500 IU SQ + FSH 450 IU SQ.

For the control arm, the standard hCG dose will be given based on the estradiol (E2) level. If the E2 level is less than 3,500 pg/ml then we will trigger with 10,000 IU of hCG. If the E2 level is more than 3,500 pg/ml but less than 5,000 pg/ml then we will trigger with 5,000 IU.

Interventions to prevent OHSS in high risk patients:

Any patients in either arm with an E2 serum level >5,000 pg/ml on the day of expected trigger administration will be excluded from the study. These patients will be individually assessed by their primary physician. Their primary physician will decide the safest trigger option based on the patient's risk of OHSS. From our own clinical experience, we expect that <5% of subjects will have an E2 serum level of >5,000 pg/ml and be excluded.

The hCG and FSH trigger shots for each patient will be prepared by one unblinded physician the same day the patient will administer the medications. The subjects will self-administer the ovulation trigger at the designated time given by the primary physician.

The oocyte retrieval will be performed 36 hours after the oocyte maturation trigger. All egg retrievals will be performed using transvaginal ultrasound and the associated needle guide in the standard fashion. Both the physician and the laboratory personnel will be blinded to the study. All visible follicles will be aspirated. The first follicle from each ovary on every patient will be aspirated and the system (needle and tubing) will be flushed into a separate tube prior to aspirating the remaining follicles so that direct correlation of follicular size to oocyte recovery maturation, and embryo development can be separately assessed. Additionally, the follicular fluid from the first aspirate will be collected for future hormone assays. Oocyte stripping will be performed under the standard protocol. The status of oocyte maturation at the time of stripping (approximately 38-40 hours after hCG administration) and at the end of the intracytoplasmic sperm injection (ICSI) procedure (approximately 40-42 hours after hCG administration) will be recorded. Fertilization will be assessed 16-19 hours after insemination. The embryos will be transferred to growth media and cultured with standard protocols.

Subjects will return 12 hours after trigger (T+1), at oocyte retrieval (T+2), and 5 days after trigger (T+5) to assess serum levels of estradiol, progesterone, hCG, FSH, LH, and vascular endothelial growth factor (VEGF), as appropriate, based on the study visit day.

To assess the incidence of OHSS, patients will be evaluated objectively by a change in the abdominal circumference as well as subjectively by clinical symptomatology based on patient's bloating symptoms.

Prior to starting the stimulation, the abdominal circumference (C) and body weight (BW) will also be measured in centimeters at the baseline ultrasound visit (C baseline, BW baseline). Five days after the oocyte retrieval the abdominal circumference and body weight will again be measured in centimeters (C stimulated, BW stimulated). The difference in the abdominal circumference and body weight will be calculated as follows: C baseline - C stimulated = CΔ.; BW baseline - BW stimulated = BWΔ.

The patient's clinical symptoms will be evaluated based on a bloating score reported by each patient before the trigger shot is administered and then 5 days after the oocyte retrieval will be determined. A venipuncture will also be obtained for hormone assays 5 days after oocyte retrieval.

Patients diagnosed with OHSS will be managed by a physician as clinically indicated. The number of follow-up clinic visits and hospitalizations secondary to symptoms of OHSS will be recorded.

ELIGIBILITY:
Inclusion Criteria: The target population includes couples undergoing IVF. All eligible couples will be asked to join the study. Study participants will be recruited from the Reproductive Endocrinology Clinic at University of California at San Francisco Center for Reproductive Health. Patients receiving any type of stimulation protocol for IVF will be offered participation in the study.

Exclusion Criteria:

* Age >41 years old
* Antral Follicle Count (AFC; 2-10 mm) < 8
* Body Mass Index > 30 kg/m2
* History of ≥ 2 prior canceled IVF cycles secondary to poor response
* Diagnosis of cancer
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow-up, or interpretation of study results
* Undergoing embryo co-culture
* Use of any of the following medications: Growth Hormone, Sildenafil, or Aspirin (except if being used for hypercoagulable state)
* Severe male factor infertility diagnosis. Male factor infertility diagnosis should be cleared for eligibility by the PI based on previous patient history of fertilization outcomes and/or expected fertilization outcomes of the cause of male factor infertility based on known scientific data.
* Ovulation trigger less than or greater than 36 hours to oocyte retrieval
* Serum estradiol level >5,000 pg/ml on the day of expected trigger due to high risk of OHSS

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Rosen, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California at San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Lamb JD, Shen S, McCulloch C, Jalalian L, Cedars MI, Rosen MP. Follicle-stimulating hormone administered at the time of human chorionic gonadotropin trigger improves oocyte developmental competence in in vitro fertilization cycles: a randomized, double-blind, placebo-controlled trial. Fertil Steril. 2011 Apr;95(5):1655-60. doi: 10.1016/j.fertnstert.2011.01.019. PMID 21315341
- [Background] Navot D, Bergh PA, Laufer N. Ovarian hyperstimulation syndrome in novel reproductive technologies: prevention and treatment. Fertil Steril. 1992 Aug;58(2):249-61. doi: 10.1016/s0015-0282(16)55188-7. PMID 1633889
- [Background] Klemetti R, Sevon T, Gissler M, Hemminki E. Complications of IVF and ovulation induction. Hum Reprod. 2005 Dec;20(12):3293-300. doi: 10.1093/humrep/dei253. Epub 2005 Aug 26. PMID 16126753
- [Background] McClure N, Healy DL, Rogers PA, Sullivan J, Beaton L, Haning RV Jr, Connolly DT, Robertson DM. Vascular endothelial growth factor as capillary permeability agent in ovarian hyperstimulation syndrome. Lancet. 1994 Jul 23;344(8917):235-6. doi: 10.1016/s0140-6736(94)93001-5. PMID 7913160
- [Background] Kashyap S, Parker K, Cedars MI, Rosenwaks Z. Ovarian hyperstimulation syndrome prevention strategies: reducing the human chorionic gonadotropin trigger dose. Semin Reprod Med. 2010 Nov;28(6):475-85. doi: 10.1055/s-0030-1265674. Epub 2010 Nov 16. PMID 21082506
- [Background] Tsoumpou I, Muglu J, Gelbaya TA, Nardo LG. Symposium: Update on prediction and management of OHSS. Optimal dose of HCG for final oocyte maturation in IVF cycles: absence of evidence? Reprod Biomed Online. 2009 Jul;19(1):52-8. doi: 10.1016/s1472-6483(10)60045-4. PMID 19573290
- [Background] Schmidt DW, Maier DB, Nulsen JC, Benadiva CA. Reducing the dose of human chorionic gonadotropin in high responders does not affect the outcomes of in vitro fertilization. Fertil Steril. 2004 Oct;82(4):841-6. doi: 10.1016/j.fertnstert.2004.03.055. PMID 15482757
- [Background] Kolibianakis EM, Papanikolaou EG, Tournaye H, Camus M, Van Steirteghem AC, Devroey P. Triggering final oocyte maturation using different doses of human chorionic gonadotropin: a randomized pilot study in patients with polycystic ovary syndrome treated with gonadotropin-releasing hormone antagonists and recombinant follicle-stimulating hormone. Fertil Steril. 2007 Nov;88(5):1382-8. doi: 10.1016/j.fertnstert.2006.12.058. Epub 2007 Apr 18. PMID 17445806
- [Background] Chen X, Chen SL, He YX, Ye DS. Minimum dose of hCG to trigger final oocyte maturation and prevent OHSS in a long GnRHa protocol. J Huazhong Univ Sci Technolog Med Sci. 2013 Feb;33(1):133-136. doi: 10.1007/s11596-013-1085-z. Epub 2013 Feb 8. PMID 23392722
- [Background] Zelinski-Wooten MB, Hutchison JS, Hess DL, Wolf DP, Stouffer RL. A bolus of recombinant human follicle stimulating hormone at midcycle induces periovulatory events following multiple follicular development in macaques. Hum Reprod. 1998 Mar;13(3):554-60. doi: 10.1093/humrep/13.3.554. PMID 9572409
- [Background] Bianchi V, Dal Prato L, Maccolini A, Mazzone S, Borini A. Inadvertent recombinant human follicle stimulating hormone bolus instead of human chorionic gonadotrophin leads to the retrieval of competent oocytes in IVF program. Fertil Steril. 2009 Nov;92(5):1747.e1-3. doi: 10.1016/j.fertnstert.2009.07.998. Epub 2009 Sep 3. PMID 19732874
- [Background] Wikland M, Borg J, Forsberg AS, Jakobsson AH, Svalander P, Waldenstrom U. Human chorionic gonadotrophin self-administered by the subcutaneous route to induce oocyte maturation in an in-vitro fertilization and embryo transfer programme. Hum Reprod. 1995 Jul;10(7):1667-70. doi: 10.1093/oxfordjournals.humrep.a136152. PMID 8582958
- [Background] Hoff JD, Quigley ME, Yen SS. Hormonal dynamics at midcycle: a reevaluation. J Clin Endocrinol Metab. 1983 Oct;57(4):792-6. doi: 10.1210/jcem-57-4-792. PMID 6411753
- [Background] Golan A, Ron-el R, Herman A, Soffer Y, Weinraub Z, Caspi E. Ovarian hyperstimulation syndrome: an update review. Obstet Gynecol Surv. 1989 Jun;44(6):430-40. doi: 10.1097/00006254-198906000-00004. No abstract available. PMID 2660037
- [Background] Egbase PE, Sharhan MA, Masangcay M, Egbase E. Follicle stimulating hormone (FSH) administer with trigger dose human chorionic gonadotropin (hCG) completely prevents ovarian hyperstimulation (OHSS): Randomised controlled study. [Abstract] Fertil Steril 2011; 96(3): S20.
- [Derived] Anaya Y, Cakmak H, Mata DA, Letourneau J, Zhang L, Lenhart N, Juarez-Hernandez F, Jalalian L, Cedars MI, Rosen M. Triggering with 1,500 IU of human chorionic gonadotropin plus follicle-stimulating hormone compared to a standard human chorionic gonadotropin trigger dose for oocyte competence in in vitro fertilization cycles: a randomized, double-blinded, controlled noninferiority trial. Fertil Steril. 2022 Aug;118(2):266-278. doi: 10.1016/j.fertnstert.2022.05.006. Epub 2022 Jun 12. PMID 35705380

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixteen patients were excluded prior to starting their IVF cycle (i.e., 9 withdrew and 7 became spontaneously pregnant), and 15 were excluded prior to randomization due to cycle cancellation for poor response or having an E2 >5,000 pg/ml on T+0.
Period: Overall Study
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Started | 54 | 51
Completed | 54 (Four participants receiving the study trigger deviated from protocol. One patient was randomized before her E2 resulted >5,000 pg/ml. Another elected to convert to intrauterine insemination while another underwent oocyte cryopreservation as their male partner was unable to produce a fresh sperm sample for fertilization. The 4th patient inadvertently spilled a portion of the trigger prior to injection. Since her post-trigger hCG was <18 IU/L, she was unblinded and re-triggered with 10,000 IU hCG.) | 51 (Two participants that received the standard trigger requested exclusionary embryo co-culture to be added post-trigger.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Dose hCG Plus FSH Co-trigger: On the day of ovulation trigger the patient will receive Low dose hCG 1,500 IU subcutaneously plus FSH 450 IU co-trigger subcutaneously
- Standard Dose of hCG Alone: On the day of ovulation trigger the patient will receive standard dose of hCG 10,000 or 5,000 IU subcutaneously.
- Total: Total of all reporting groups
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone | Total
Number analyzed (Participants) | 54 | 51 | 105
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37.5 [34.3 to 40.0] | 37.0 [35.0 to 39.0] | 37.0 [34.5 to 40.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 51 | 105
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 22.8 [21.4 to 25.6] | 22.8 [21.2 to 25.4] | 22.8 [21.3 to 25.6]
Baseline antral follicle count (AFC) [Median (Inter-Quartile Range); unit: follicles] | 14.5 [11.0 to 19.0] | 15.0 [11.5 to 18.0] | 15.0 [11.0 to 18.0]
Number of prior IVF attempts [Median (Inter-Quartile Range); unit: IVF cycles] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
Infertility Diagnosis [Count of Participants; unit: Participants]
  Unexplained | 23 | 24 | 47
  Male factor | 7 | 11 | 18
  Tubal factor | 3 | 2 | 5
  Other | 21 | 14 | 35
Total dose of gonadotropins [Median (Inter-Quartile Range); unit: International Units (IU)] — Total dose of gonadotropins used per cycle
  International Units (IU) | 3750.0 [2700.0 to 4125.0] | 3375.0 [2700.0 to 3788.0] | 3525.0 [2700.0 to 4125.0]
Length of stimulation [Median (Inter-Quartile Range); unit: days] — Length of IVF stimulation cycle in days
  days | 11.0 [10.0 to 12.0] | 11.0 [10.0 to 12.0] | 11.0 [10.0 to 12.0]
Number of follicles on T+0 [Median (Inter-Quartile Range); unit: follicles] — Number of follicles counted on day of trigger
  follicles | 18.5 [14.0 to 22.0] | 17.0 [14.0 to 23.5] | 18.0 [14.0 to 23.0]
Serum estradiol on T+0 [Median (Inter-Quartile Range); unit: pg/ml] — Serum estradiol level on day of trigger
  pg/ml | 2871.0 [2050.8 to 3869.2] | 2911.0 [2330.0 to 3638.0] | 2883.0 [2081.5 to 3779.5]

OUTCOME MEASURES:

1. Primary Outcome: Total Fertilization Proportion (i.e. Total Competent Proportion)
Description: The number of fertilized oocytes (2-pronuclei) after standard in vitro fertilization or intra-cytoplasmic sperm injection divided by the total number of oocytes retrieved as a measure of oocyte competence.
Time Frame: 2 days
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 54 | 51
ratio | 0.59 (0.029) | 0.65 (0.024)
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; The alternative trigger will be considered non-inferior to the standard hCG trigger if it is at least 80% as effective at inducing oocyte competence. Considering a cluster size of 15 oocytes and an estimated intra-cluster correlation of 0.1, we calculated that approximately 50 participants were needed in each study arm when the non-inferiority difference is -0.1 (i.e. 20% of 0.5 total competent proportion) with a power of 0.8 and a one-sided alpha of 0.05; Test type: Non-Inferiority — For the non-inferiority hypothesis testing of the primary outcome, a one-sided 95% CI was constructed for the relative risk. The alternative trigger will be considered non-inferior to the standard trigger if the lower bound of the one-sided CI of the relative risk is not less than 0.8 (i.e. risk reduction limit of 20%); log-binomial regression with GEE — Using the standard trigger as the reference, the relative risk (i.e. risk ratio) (RR) with 95% confidence interval (CI) for the probability of the outcome was calculated using log-binomial regression models with application of GEE; Risk Ratio (RR) = 0.91, 95% CI 1-sided [lower limit 0.83] — The numerator was the probability of the outcome with the alternative trigger, and the denominator was the probability of the outcome with the standard trigger

2. Secondary Outcome: Number of Oocytes Retrieved
Description: The total number of oocytes recovered at the oocyte retrieval.
Time Frame: 1 day
Population: No outcome data for 1 participant that elected to convert to intrauterine insemination after trigger
Measure: Mean (Standard Error); unit: oocytes
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 53 | 51
oocytes | 13.6 (0.84) | 16.1 (1.01)
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; The null hypothesis was that there would be no difference in number of oocytes retrieved between the patients triggered with low dose hCG plus FSH co-trigger and the standard hCG trigger; Test type: Superiority; p = 0.06, generalized linear model with log link — The statistical significance was based on a two-sided alpha of 0.05; Comparison was done using generalized linear modeling with log link function; Risk Ratio (RR) = 0.85, 95% CI 2-sided [0.71 to 1.01] — The numerator was the outcome with the alternative trigger, and the denominator was the outcome with the standard trigger

3. Secondary Outcome: Number of MII Oocytes
Description: The number of metaphase 2 oocytes (MII) recovered which can only be calculated in patients that underwent intracytoplasmic sperm injection.
Time Frame: 1 day
Population: This parameter can only be calculated in patients that underwent oocyte stripping to undergo intracytoplasmic sperm injection for fertilization method.
Measure: Mean (Standard Error); unit: MII oocytes
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 39 | 44
MII oocytes | 10.8 (0.74) | 12.5 (0.81)
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; The null hypothesis was that there would be no difference in the number of MII oocytes retrieved between the patients triggered with low dose hCG plus FSH co-trigger and the standard hCG trigger; Test type: Superiority; p = 0.13, generalized linear model with log link — The statistical significance was based on a two-sided alpha of 0.05; Comparison was done using generalized linear modeling with log link function; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.72 to 1.04] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Total Oocyte Maturity Rate
Description: Oocyte maturity rate was determined by the number of meta phase 2 (MII) oocytes divided by the number of oocytes retrieved. This outcome was only assessed in patients undergoing intracytoplasmic sperm injection (ICSI).
Time Frame: 1 day
Population: as for outcome 3
Measure: Mean (Standard Error); unit: ratio of MII oocytes
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 39 | 44
ratio of MII oocytes | 0.75 (0.021) | 0.77 (0.020)
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; The null hypothesis was that there would be no difference in oocyte maturity rate retrieved between the patients triggered with low dose hCG plus FSH co-trigger and the standard hCG trigger; Test type: Superiority; p = 0.47, log-binomial regression with GEE — The statistical significance was based on a two-sided alpha of 0.05; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.90 to 1.05] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Mature Oocyte Recovery Proportion
Description: Mature oocyte recovery proportion is defined as the number of MIIs divided by the total number of follicles greater or equal to 13mm in size on trigger day.
Time Frame: 1 day
Population: as for outcome 3
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 39 | 44
ratio | 0.81 (0.032) | 0.92 (0.018)
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p = 0.01, log-binomial regression with GEE — The statistical significance was based on a two-sided alpha of 0.05; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.76 to 0.97] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: ICSI Fertilization Rate
Description: ICSI fertilization rate was determined by the number of 2 pro-nuclei (2PN) divided by the number of MII oocytes. This was only assessed in patients undergoing ICSI.
Time Frame: 2 days
Population: This parameter can only be calculated in patients that were undergoing intracytoplasmic sperm injection for fertilization method. One participant the low dose hCG plus FSH co-trigger arm was not included in the analysis as they underwent oocyte cryopreservation instead as the male partner was unable to produce fresh sperm sample to fertilize the oocytes.
Measure: Mean (Standard Error); unit: ratio of fertilized oocytes
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 38 | 44
ratio of fertilized oocytes | 0.80 (0.032) | 0.80 (0.024)
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; The null hypothesis was that there would be no difference in ICSI fertilization rate retrieved between the patients triggered with low dose hCG plus FSH co-trigger and the standard hCG trigger; Test type: Superiority; p = 0.95, log-binomial regression with GEE — The statistical significance was based on a two-sided alpha of 0.05; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.90 to 1.10] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: High Quality Cleavage-stage Embryos
Description: Good quality embryo development was compared between trigger groups by calculating the ratio of good quality embryos to the total number of cleavage-stage embryos. A good quality cleavage-stage embryo was defined by having a cell number of 7 to 10 and <10% of cell fragmentation based on a modified Veeck's grading system.
Time Frame: 4 days
Population: No outcome data for 3 participants: 1) participant that elected to convert to intrauterine insemination after trigger; 2) participant that underwent oocyte cryopreservation due to male partner being unable to produce fresh sperm sample for fertilization; 3) cleavage-stage embryo quality was inadvertently not documented by the staff embryologist in one participant
Measure: Mean (Standard Error); unit: ratio of good quality embryos
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 51 | 51
ratio of good quality embryos | 0.59 (0.043) | 0.62 (0.027)
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; The null hypothesis was that there would be no difference in the percentage of high quality cleavage-stage embryos between the patients triggered with low dose hCG plus FSH co-trigger and the standard hCG trigger; Test type: Superiority; p = 0.52, log-binomial regression with GEE — The statistical significance was based on a two-sided alpha of 0.05; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.81 to 1.12] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: High Quality Blastocyst Embryos
Description: A high quality blastocyst was defined as grade 3 or higher expansion plus inner cell mass and trophectoderm grading of A or B based on Gardner's criteria. The number describes the degree of embryo expansion on a scale from 1-6. As the embryo expands, the degree of expansion increases. The first letter indicates on a scale from A to C (A being the highest) the quality of the inner cell mass. The second letter is also on a scale from A to C (A being the highest) and indicates the quality of the trophectoderm.
Time Frame: 6 days
Measure: Mean (Standard Error); unit: ratio of good quality embryos
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 35 | 40
ratio of good quality embryos | 0.67 (0.044) | 0.68 (0.035)
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p = 0.87, log-binomial regression with GEE — The statistical significance was based on a two-sided alpha of 0.05; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.84 to 1.16] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Livebirth Rate From All Fresh Transfers
Description: Livebirth rate (LBR) was defined as a liveborn at the time of the analysis. Pregnancy outcomes were calculated for all fresh transfers.
Time Frame: 10 months
Population: Only patients that underwent a fresh embryo transfer can be included in this analysis. Not all participants underwent fresh embryo transfers.
Measure: Number; unit: live births
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 32 | 28
live births | 15 | 13
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; The null hypothesis was that there would be no difference in livebirths in fresh transfers between the patients triggered with low dose hCG plus FSH co-trigger and the standard hCG trigger; Test type: Superiority; p = 1.0, Fisher Exact — The statistical significance was based on a two-sided alpha of 0.05; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.59 to 1.74] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Bloating Score
Description: Change in bloating scores from day of baseline ultrasound to post-trigger day 5.
  The patient's clinical symptoms will be evaluated based on a bloating score reported by each patient on the day of ovulation trigger and then 5 days after the oocyte retrieval will be determined. The bloating score will range on a scale from 0-5. The number describes the degree of bloating and will increase as the degree of bloating increases. The bloating score will be determined as follows:
  0 - No bloating
  1. - Mild bloating. Able to continue daily activities without discomfort.
  2. - Mild to moderate bloating. Able to continue daily activities but with mild discomfort.
  3. - Moderate bloating. Able to continue daily activities but with moderate discomfort.
  4. - Moderate to severe bloating. Difficulty performing daily activities.
  5. - Severe bloating. Abdomen feels very tense and unable to perform daily activities.
Time Frame: about 16 days (varies by subject), accounts for the median length of IVF stimulation in this study being 11 days from baseline to 5 days post trigger
Population: Only patients that answered this question on the study questionnaire could be included in this analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 48 | 47
score on a scale | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; The null hypothesis was that there would be no difference in the change in bloating scores from day of baseline ultrasound to post-trigger day 5 between the patients triggered with low dose hCG plus FSH co-trigger and the standard hCG trigger; Test type: Superiority; p = 0.98, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Abdominal Circumference
Description: Change in abdominal circumference (in centimeters) from day of baseline ultrasound to post-trigger day 5.
Time Frame: as for outcome 10
Population: Only patients that had their abdominal circumference measured on both day of baseline ultrasound and post-trigger day 5 could be included in this analysis.
Measure: Median (Inter-Quartile Range); unit: centimeters
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 48 | 48
centimeters | 0.38 [-3.25 to 2.88] | 1.00 [-2.00 to 4.88]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; The null hypothesis was that there would be no difference in the change in abdominal circumference from day of baseline ultrasound to post-trigger day 5 between the patients triggered with low dose hCG plus FSH co-trigger and the standard hCG trigger; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Body Weight
Description: Change in body weight from day of baseline ultrasound to post-trigger day 5.
Time Frame: as for outcome 10
Population: Only patients that had their body weight measured on both day of baseline ultrasound and post-trigger day 5 could be included in this analysis.
Measure: Median (Inter-Quartile Range); unit: difference in kilograms
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 49 | 50
difference in kilograms | 0.10 [-0.35 to 0.70] | 0.05 [-0.53 to 0.53]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; The null hypothesis was that there would be no difference in the change in body weight from day of baseline ultrasound to post-trigger day 5 between the patients triggered with low dose hCG plus FSH co-trigger and the standard hCG trigger; Test type: Superiority; p = 0.41, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Serum hCG T+1
Description: Blood samples were collected about 12 hours after trigger (T+1) to assess the serum concentration of human chorionic gonadotropin (hCG).
Time Frame: 1 day
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: IU/L
Groups:
- Standard Dose of hCG Alone: On the day of ovulation trigger the patient will receive standard dose of 10,000 IU hCG subcutaneously.
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
IU/L | 56.1 [39.0 to 65.6] | 267.4 [227.3 to 322.3]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

14. Secondary Outcome: Serum FSH T+1
Description: Blood samples were collected about 12 hours after trigger (T+1) to assess the serum concentration of follicle stimulating hormone (FSH).
Time Frame: 1 day
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: mIU/ml
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
mIU/ml | 29.6 [24.0 to 34.3] | 19.0 [14.2 to 22.9]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

15. Secondary Outcome: Serum P4 on T+1
Description: Blood samples were collected about 12 hours after trigger (T+1) to assess the serum concentration of Progesterone (P4).
Time Frame: 1 day
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
ng/ml | 6.1 [4.2 to 8.5] | 7.0 [5.4 to 11.1]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

16. Secondary Outcome: Serum E2 on T+1
Description: Blood samples were collected about 12 hours after trigger (T+1) to assess the serum concentration of estradiol (E2).
Time Frame: 1 day
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
pg/ml | 4010 [2612 to 4919] | 2763 [1994 to 3341]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

17. Secondary Outcome: Serum LH on T+1
Description: Blood samples were collected about 12 hours after trigger (T+1) to assess the serum concentration of luteinizing hormone (LH).
Time Frame: 1 day
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: mIU/ml
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
mIU/ml | 1.75 [1.04 to 3.94] | 1.70 [0.66 to 3.96]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p = 0.67, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

18. Secondary Outcome: Serum hCG on T+2
Description: Blood samples were collected about 2 days after trigger (T+2) to assess the serum concentration of human chorionic gonadotropin (hCG).
Time Frame: 2 days
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
IU/L | 52.6 [40.6 to 62.0] | 271.3 [218.3 to 318.9]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

19. Secondary Outcome: Serum FSH on T+2
Description: Blood samples were collected 2 days after trigger (T+2) to assess the serum concentration of follicle stimulating hormone (FSH).
Time Frame: 2 days
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: mIU/ml
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
mIU/ml | 20.5 [16.1 to 24.9] | 12.0 [9.7 to 14.1]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

20. Secondary Outcome: Serum P4 on T+2
Description: Blood samples were collected 2 days after trigger (T+2) to assess the serum concentration of progesterone (P4).
Time Frame: 2 days
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
ng/ml | 10.7 [7.4 to 13.9] | 10.0 [6.9 to 13.9]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

21. Secondary Outcome: Serum E2 on T+2
Description: Blood samples were collected 2 days after trigger (T+2) to assess the serum concentration of estradiol (E2).
Time Frame: 2 days
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
pg/ml | 1773 [1304 to 2112] | 955 [802 to 1205]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

22. Secondary Outcome: Serum HCG on T+5
Description: Blood samples were collected 5 days after trigger (T+5) to assess the serum concentration of human chorionic gonadotropin (hCG).
Time Frame: 5 days
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
IU/L | 9.5 [5.9 to 12.5] | 52.1 [44.4 to 77.6]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

23. Secondary Outcome: Serum FSH on T+5
Description: Blood samples were collected 5 days after trigger (T+5) to assess the serum concentration of follicle stimulating hormone (FSH).
Time Frame: 5 days
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: mIU/ml
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
mIU/ml | 5.1 [3.9 to 7.0] | 3.2 [2.8 to 4.0]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

24. Secondary Outcome: Serum LH on T+5
Description: Blood samples were collected about 5 days after trigger (T+5) to assess the serum concentration of luteinizing hormone (LH).
Time Frame: 5 days
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: mIU/ml
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
mIU/ml | 0.65 [0.60 to 1.08] | 0.61 [0.55 to 0.91]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

25. Secondary Outcome: Follicular hCG
Description: Follicular fluid was individually aspirated at oocyte retrieval from the lead follicle in each ovary using a single lumen needle. The mean concentration between right and left follicles collected was compared to assess the follicular concentration of human chorionic gonadotropin (hCG).
Time Frame: 2 days
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
IU/L | 11.6 [7.0 to 17.5] | 135.3 [100.5 to 165.8]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

26. Secondary Outcome: Follicular FSH
Description: Follicular fluid was individually aspirated at oocyte retrieval from the lead follicle in each ovary using a single lumen needle. The mean concentration between right and left follicles collected was compared to assess the follicular concentration of follicle stimulating hormone (FSH).
Time Frame: 2 days
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: mIU/ml
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
mIU/ml | 13.1 [10.0 to 15.4] | 9.2 [6.7 to 11.0]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

27. Secondary Outcome: Follicular P4
Description: Follicular fluid was individually aspirated at oocyte retrieval from the lead follicle in each ovary using a single lumen needle. The mean concentration between right and left follicles collected was compared to assess the follicular concentration of progesterone (P4).
Time Frame: 2 days
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
ng/ml | 26095 [22445 to 38525] | 28758 [23015 to 37838]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

28. Secondary Outcome: Follicular E2
Description: Follicular fluid was individually aspirated at oocyte retrieval from the lead follicle in each ovary using a single lumen needle. The mean concentration between right and left follicles collected was compared to assess the follicular concentration of estradiol (E2).
Time Frame: 2 days
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
pg/ml | 842.2 [576.5 to 1321.1] | 672.7 [456.1 to 1021.2]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

29. Secondary Outcome: Follicular VEGF
Description: Follicular fluid was individually aspirated at oocyte retrieval from the lead follicle in each ovary using a single lumen needle. The mean concentration between right and left follicles collected was compared to assess the follicular concentration of vascular endothelial growth factor (VEGF).
Time Frame: 2 days
Population: Only comparisons to the standard 10,000 IU hCG trigger dose are presented using the per-protocol study population.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
Number analyzed (Participants) | 50 | 35
pg/ml | 3436 [2289 to 4352] | 3470 [2596 to 4522]
Statistical Analysis 1: Comparison: Low Dose hCG Plus FSH Co-trigger vs Standard Dose of hCG Alone; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney) — The statistical significance was based on a two-sided alpha of 0.05

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Low Dose hCG Plus FSH Co-trigger | Standard Dose of hCG Alone
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/54 | 1/51
Other Adverse Events (participants affected / at risk) | 0/54 | 1/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose hCG Plus FSH Co-trigger (N=54) | Standard Dose of hCG Alone (N=51)
Severe OHSS (Reproductive system and breast disorders) | 0 | 1 (1) — Severe Ovarian Hyperstimulation Syndrome (OHSS)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose hCG Plus FSH Co-trigger (N=54) | Standard Dose of hCG Alone (N=51)
Mild OHSS (Reproductive system and breast disorders) | 0 | 1 (1) — Mild Ovarian Hyperstimulation Syndrome (OHSS)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT02310919/Prot_SAP_000.pdf